CLINICAL TRIAL: NCT03383575
Title: Targeted Therapy With the IDH2-Inhibitor Enasidenib (AG221) for High-Risk IDH2-Mutant Myelodysplastic Syndrome
Brief Title: Azacitidine and Enasidenib in Treating Patients With IDH2-Mutant Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0981; NCI-2018-00987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0981 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Blasts 20-30 Percent of Bone Marrow Nucleated Cells; Chronic Myelomonocytic Leukemia; IDH2 Gene Mutation; Myelodysplastic Syndrome With Excess Blasts; Recurrent High Risk Myelodysplastic Syndrome; Refractory High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts | interventions — Azacitidine; enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (enasidenib, azacitidine) (Experimental): Patients who are HMA-naive receive enasidenib PO QD on days 1-28 and azacitidine IV over 30-60 minutes or SC on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Enasidenib; Other: Quality-of-Life Assessment
- Arm II (enasidenib) (Experimental): Patients relapsed and/or refractory to HMA therapy receive enasidenib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enasidenib; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Arm I (enasidenib, azacitidine)
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the side effects and how well azacitidine and enasidenib work in treating patients with IDH2-mutant myelodysplastic syndrome. Azacitidine and enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of enasidenib alone, and enasidenib in combination with azacitidine (AZA), for patients with isocitrate dehydrogenase 2 (IDH2) mutated myelodysplastic syndrome (MDS).

II. To assess the efficacy of the combination of enasidenib + azacitidine in hypomethylating agent (HMA) naive subjects with IDH2-mutated MDS, and to assess the efficacy of enasidenib single-agent in subjects with IDH2-mutated MDS who are relapsed/refractory to HMA therapy.

SECONDARY OBJECTIVES:

I. To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance including evaluation of IDH2 variant allele fraction (VAF) levels during treatment and presence of co-occurring mutations.

II. To assess overall survival, event-free survival and duration of response of enasidenib alone, and enasidenib in combination with azacitidine.

EXPLORATORY OBJECTIVES:

I. To assess changes in cellular differentiation and changes in deoxyribonucleic acid (DNA) methylation profiles in IDH2-mutated MDS treated with enasidenib alone and with enasidenib + azacitidine.

II. To evaluate quality of life (QOL) using an MDS-specific measure.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients who are HMA-naive receive enasidenib orally (PO) once daily (QD) on days 1-28 and azacitidine intravenously (IV) oveer 30-60 minutes or subcutaneously (SC) on days 1-7. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients relapsed and/or refractory to HMA therapy receive enasidenib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent must be obtained prior to any study specific procedures
* Subjects with a histologically confirmed diagnosis of MDS, including both MDS and refractory anemia with excess blasts in transformation (RAEB-T) (acute myeloid leukemia [AML] with 20-30% blasts and multilineage dysplasia by French-American-British [FAB] criteria) by World Health Organization (WHO), and chronic myelomonocytic leukemia (CMML) are eligible
* Subjects must have an IDH2 gene mutation (IDH2-R140 or R172) as determined by local laboratory result
* (Arm A only): Subject must be hypomethylating agent naive (i.e. prior azacitidine, decitabine, SGI-110 is exclusionary). Receipt of other MDS-directed therapy such as lenalidomide is allowed
* (Arm A only): Subjects with high-risk MDS (i.e. International Prostate Symptom Score [IPSS] intermediate-2 or high-risk; or revised [R]-IPSS high or very-high risk). Patients with intermediate-1 risk by IPSS or intermediate risk by R-IPSS with high-risk molecular features including TP53, ASXL1, EZH2, and/or RUNX1 mutations are also eligible
* (Arm B only): Subject must be relapsed or refractory to prior hypomethylating agent therapy, defined as prior receipt of 6 cycles of HMA therapy with failure to attain a response, or relapse after prior response to HMA therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Serum bilirubin =< 2 x the upper limit of normal (ULN) (except for patients with Gilbert's disease)
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 3 x the laboratory ULN
* Serum creatinine =< 2 x the ULN
* Able to understand and voluntarily sign a written informed consent, and willing and able to comply with protocol requirements
* Resolution of all clinically significant treatment-related, non-hematological toxicities, except alopecia, from any previous cancer therapy to =< grade 1 prior to the first dose of study treatment
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days of the first dose of study drug and agree to use dual methods of contraception during the study and for a minimum of 3 months following the last dose of study drug. Post-menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from these requirements. Male patients must use an effective barrier method of contraception during the study and for a minimum of 3 months following the last dose of study drug if sexually active with a female of childbearing potential

Exclusion Criteria:

* Any prior or coexisting medical condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study
* Subject has received a prior targeted IDH2 inhibitor
* Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures
* Active uncontrolled infection at study enrollment including known diagnosis of human immunodeficiency virus or chronic active hepatitis B or C infection
* Clinically significant gastrointestinal conditions or disorders that may interfere with study drug absorption, including prior gastrectomy
* Patients with known active central nervous system (CNS) disease, including leptomeningeal involvement
* Impaired cardiac function, uncontrolled cardiac arrhythmia, or clinically significant cardiac disease including the following: a) New York Heart Association grade III or IV congestive heart failure, b) myocardial infarction within the last 6 months
* Subjects with a corrected QT (QTc) > 480 ms (QTc > 510 msec for subjects with a bundle branch block at baseline
* Nursing or pregnant women
* Subjects with known hypersensitivity to study drugs or their excipients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Will use the Bayesian method by Thall, Simon and Estey for toxicity monitoring. For purpose of toxicity monitoring, toxicity is defined as any grade 3 or higher treatment related-toxicities by Common Terminology Criteria for Adverse Events criteria.
Overall response rate | Up to 3 years
  Defined as complete response (CR), partial response, and marrow CR assessed by International Working Group criteria. Will be estimated along with the 90% credible interval.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of EFS. Log-rank tests will be used to compare among subgroups of patients in terms of EFS.
Overall survival (OS) | Up to 3 years
  The Kaplan-Meier method will be used to estimate the probabilities of OS. Log-rank tests will be used to compare among subgroups of patients in terms of OS.
Anti-tumor activity | Up to 3 years
  Will be summarized graphically and with descriptive statistics.
Pharmadynamics (PDn) markers | Up to 3 years
  PDn markers will be summarized graphically and with descriptive statistics.
Drug exposure levels | Up to 3 years
  Will be summarized graphically and with descriptive statistics.

OTHER OUTCOMES:
Biomarkers analysis | Up to 3 years
  The association between molecular and cellular markers and overall response and/or resistance will be assessed through logistic regression analyses. Paired t-test or Wilcoxon signed rank test will be used to assess the marker change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] DiNardo CD, Venugopal S, Lachowiez C, Takahashi K, Loghavi S, Montalban-Bravo G, Wang X, Carraway H, Sekeres M, Sukkur A, Hammond D, Chien K, Maiti A, Masarova L, Sasaki K, Alvarado Y, Kadia T, Short NJ, Daver N, Borthakur G, Ravandi F, Kantarjian HM, Patel B, Dezern A, Roboz G, Garcia-Manero G. Targeted therapy with the mutant IDH2 inhibitor enasidenib for high-risk IDH2-mutant myelodysplastic syndrome. Blood Adv. 2023 Jun 13;7(11):2378-2387. doi: 10.1182/bloodadvances.2022008378. PMID 35973199
- See also: Related Info — http://mdanderson.org